CLINICAL TRIAL: NCT05555810
Title: Suture Ligation Versus Clipping of Cystic Duct and Artery During Laparoscopic Cholecystectomy . " A Prospective Comparative Study"
Brief Title: Suture Ligation Versus Clipping of Cystic Duct and Artery During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Sayed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lclc
Record Dates: First submitted 2022-09-17; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: The investigators will secure Cystic duct and artery with traditional sutures(ligation) in a group. In the another group the cystic duct and artery will be put a clips .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture ligation of cystic duct and artery (Active Comparator): The investigators will ligate cystic duct and artery by traditional sutures during laparoscopic cholecystectomy .
  Interventions: Procedure: clipping or ligation of the cystic duct and the cystic artery in Laparoscopic cholecystectomy
- Application of clips (Active Comparator): The investigators will put a clips on the cystic duct and artery during laparoscopic cholecystectomy.
  Interventions: Procedure: clipping or ligation of the cystic duct and the cystic artery in Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: clipping or ligation of the cystic duct and the cystic artery in Laparoscopic cholecystectomy — The investigators will make a comparison between clipping and ligation of cystic duct and cystic artery during Laparoscopic cholecystectomy and trying to know advantages and disadvantages of each technique .

SUMMARY:
The investigators will compare between clipping and ligation of the cystic duct and the cystic artery in Laparoscopic cholecystectomy. This is the main question that will be discussed in the review.

DETAILED DESCRIPTION:
cholecystectomy is the second most commonly intra-abdominal operation worldwide after Appendectomy. In standard surgery ,there are increase incidence of wound infection,bleeding , discomfort and hospital stay so laparoscopic surgery has become the best choice for treatment of symptomatic and uncomplicated Gall bladder stones and hernia repair.

Once laparoscopic cholecystectomy emerged controversies persist with regard to the best method to ligate the cystic duct and artery. They may be ligated by separate and multiple ligatures by absorbable suture material, or using absorbable clips.

Suture ligation of cystic duct appeared to be more cost effective.On the other hand, the application of clips shown to have some drawbacks such as dislodgement and bile leakage and increase liability of long term clip migration which resulted in biliary stone formation or bile duct stenosis and also they are expensive .Another complication of clips that they may ulcerated through the duodenum.

Ligation takes more time than applying a clip, and it needs well training, but it is feasible, cost- effective and safe alternative method to secure cystic duct and artery in laparoscopic cholecystectomy.

The Aim of this study is to compare the two different methods; Tie versus clipping, for securing cystic duct and artery in laparoscopic cholecystectomy. In terms of efficacy and safety, and also the difference in the times of operations in both methods

ELIGIBILITY:
Inclusion Criteria:

* patients with cholecystitis admitted at Assuit University Hospital and planed for lap. cholecystectomy the period of the study

Exclusion Criteria:

* Any case not candidate for laparoscopic cholecystectomy and we must do it by open technique .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
safety and efficiency of closure of cystic duct and artery after cutting them during laparoscopic cholecystectomy | one month
  The investigators will seek to know the incidence of postoperative complications of laparoscopic cholecystectomy (as signs of biliary leakage as pain, jaundice and raised serum bilirubin level and follow up the drain inserted after doing laparoscopic cholecystectomy)
  then the investigators will make a comparison between incidence of these complication after closure of cystic duct and artery either by clipping or ligation by sutures.
  The investigators will try to know rate of advantages disadvantages of each technique also do our best to make strategies for improving efficiency and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Korany, PHD, Study Director — Assut University

REFERENCES:
- [Background] van Dijk AH, van Roessel S, de Reuver PR, Boerma D, Boermeester MA, Donkervoort SC. Systematic review of cystic duct closure techniques in relation to prevention of bile duct leakage after laparoscopic cholecystectomy. World J Gastrointest Surg. 2018 Sep 27;10(6):57-69. doi: 10.4240/wjgs.v10.i6.57. PMID 30283606
- [Background] Singal R, Sharma A, Zaman M. The Safety and Efficacy of Clipless versus Conventional Laparoscopic Cholecystectomy - our Experience in an Indian Rural Center. Maedica (Bucur). 2018 Mar;13(1):34-43. PMID 29868139